CLINICAL TRIAL: NCT03184415
Title: A Multi-Center, Randomized, Parallel, Double-Blind, Phase III Clinical Trial to Compare the Efficacy and Safety of DWC20155/DWC20156 Combination Therapy With DWC20155 or DWC20156 Monotherapy in Patients With Gastritis
Brief Title: Efficacy and Safety of DWC20155/DWC20156 Combination Therapy in Patients With Gastritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWJ1366006
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Gastritis
MeSH Terms: conditions — Gastritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DWC20155/DWC20156 Combination Therapy (Experimental)
  Interventions: Drug: DWC20155; Drug: DWC20156; Drug: placebo of DWC20155
- DWC20155 Monotherapy (Active Comparator)
  Interventions: Drug: DWC20155; Drug: placebo of DWC20155; Drug: placebo of DWC20156
- DWC20156 Monotherapy (Active Comparator)
  Interventions: Drug: DWC20156; Drug: placebo of DWC20155

INTERVENTIONS:
Drug: DWC20155 — tablet
  Arms: DWC20155 Monotherapy; DWC20155/DWC20156 Combination Therapy
Drug: DWC20156 — tablet
  Arms: DWC20155/DWC20156 Combination Therapy; DWC20156 Monotherapy
Drug: placebo of DWC20155 — tablet
Drug: placebo of DWC20156 — tablet
  Arms: DWC20155 Monotherapy

SUMMARY:
THe purpose of this study is to evaludate the Efficacy and Safety of DWC20155/DWC20156 Combination Therapy in Patients with Gastritis

ELIGIBILITY:
Inclusion Criteria:

* Male of female of at least 19 years old
* Patients diagnosed with acute or chronic gastritis by gastroscopy
* Patients with one or more erosions found by gastroscopy

Exclusion Criteria:

* Patients with peptic ulcer and gastroesophageal reflux disease
* Patients with previous gastrointestinal surgery
* Patients with history of gastrointestinal cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Improvement rates of stomach erosions by the endoscopy | At 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Daewoong pharmatceutical, Seoul, South Korea